CLINICAL TRIAL: NCT07320612
Title: Efficacy And Safety Of Azithromycin To Achieve Remissionin In Children With Steroid Sensitive Nephrotic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Ummara Subhani, Principal investigator, University of Child Health Sciences and Children's Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 08-03-2025Approved by UCHS
Record Dates: First submitted 2025-11-26; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Azithromycin; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group taking Azithromycin and Steroids (Experimental): 80 Children will be assigned group A in which children will be given Azithromycin at 10mg /kg/day Per oral along with standard course of treatment.
  Interventions: Drug: Azithromycin and steroids
- Group Taking steroids (Active Comparator): 80 Children will be assigned group B in which children will be only given standard course of steroids.
  Interventions: Drug: steroids

INTERVENTIONS:
Drug: Azithromycin and steroids — 80 children will be assigned group A and children will be given Azithromycin along with standard course of steroids.
  Other Names: Azithromycin
  Arms: Group taking Azithromycin and Steroids
Drug: steroids — 80 children will be assigned group B and will be given only standard course of treatment
  Arms: Group Taking steroids

SUMMARY:
To compare efficacy and safety of Azithromycin versus control in children with steroid sensitive nephrotic syndrome

DETAILED DESCRIPTION:
It is a randomized controlled trial. Total 160 children meeting inclusion criteria will be included in the study. Selected children will be divided into 2 groups. one group will be given Azithromycin at 10mg/kg/day (1 dose per day) for 3 days along with standard course of steroids. 2nd group will be given standard course of treatment. All patients will be followed up for 1 month and remission will be noted. All data will be collected through specially designed performa. Patient's safety and Efficacy of drug in Achieving early Remission will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Children age 2 to 14 years
* Both genders
* Children having primary nephrotic syndrome

Exclusion Criteria:

* Children with steroid resistant nephrotic syndrome
* Children with secondary causes of nephrotic syndrome
* Recent use of azithromycin during last 4 weeks
* Severe systemic infection requiring antibiotics
* Chronic liver disease Prolong QT Interval or history of cardiac arythmias

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2025-03-08 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-10-08 (Actual)

PRIMARY OUTCOMES:
Early remission. | 14 days
  This study will make an impact on understanding the effectiveness and safety of azithromycin in children regain early remission. It will be classified as either complete or partial remission. Complete remission will be indicated as negative or having trace proteinuria and will be measured with the help of early morning urine dipstick test for proteinuria for 3 consecutive days, serum albumin level of more than 2.5g/dl and resolution of edema. Partial remission will be defined as serum albumin level of more than 2.5g/dl but with persistent proteinuria. Early Remission and relapse will be presented as frequency and percentage. Both groups will be compared for early remission by chi square test.

SECONDARY OUTCOMES:
Relapse reduction | 14 days
  Lower the frequency of relapses to prevent complications and minimise exposure to drugs like steroids.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Ummara Subhani, MD, Principal Investigator — UCHS Lahore
Locations (1):
- UCHS, Lahore, Punjab Province, Pakistan